CLINICAL TRIAL: NCT00375765
Title: A Randomized, Open-label, Parallel-group Study, to Assess the Pharmocodynamic Effect on Dihydrotestosterone Regulated Gene Expression, Longitudinally and in a Dose Dependent Manner, of 0.5mg and 3.5mg Dutasteride Administered Orally Once Daily, for One Year in Men With Symptomatic Benign Prostatic Hyperplasia and During a Two Month Period Between Baseline and Radical Prostatectomy in Men With Biopsy-proven, Clinically Localized Prostate Cancer
Brief Title: Effects On Dihydrotestosterone Regulated Gene Expression In Benign Prostatic Hyperplasia Or Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104274
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Benign Prostatic Hyperplasia; Prostate Cancer
Keywords: Dutasteride; BPH; Prostate cancer; Gene expression; PSA
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Neoplasms | interventions — Dutasteride

INTERVENTIONS:
Drug: Dutasteride

SUMMARY:
Dutasteride is used in the treatment of benign prostate enlargement (BPH).It inhibits conversion of testosterone (T) into the more potent dihydrotestosterone (DHT) to stop prostate (and possibly prostate cancer) growth. DHT regulates the expression of certain genes in the prostate. The pharmacodynamics of DHT reduction in the prostate were never investigated until now, as every measurement would require prostate tissue retrieval, which is medically and ethically unacceptable. A recently developed test is able to quantitatively measure gene expression in prostate-borne cells, in urine sediments after prostate massage. By measuring this gene expression in patients using dutasteride, it has become possible to assess the pharmacodynamics of gene expression reduction, which is representative for the pharmacodynamics of DHT reduction. Repeated prostate tissue sampling has therefore become unnecessary. This newly gained knowledge will lead to a better understanding of the action of dutasteride and will possibly help improve treatment of symptomatic BPH (Benign Prostatic Hyperplasia) and PrCa (Prostate Cancer)in the future.

DETAILED DESCRIPTION:
A randomized, open-label, parallel-group pilot study, to assess the pharmacodynamic effect on dihydrotestosterone regulated gene expression, longitudinally and in a dose dependent manner, of 0.5mg or 3.5mg dutasteride administered orally once daily, for three months in men with symptomatic benign prostatic hyperplasia or during the period between baseline and radical prostatectomy in men with biopsy-proven, clinically localized prostate cancer.

ELIGIBILITY:
Inclusion criteria:

* Symptomatic BPH, or:

Biopsy proven, localised (cT1 or cT2) prostate cancer scheduled for radical operation

* Able to swallow oral medication

Exclusion criteria:

* Inability to void spontaneously (eg. dependence on catheter etc.)
* History of (prior) prostate cancer Previous prostatic surgery

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Relative change in PSA(Prostate-specific antigen)expression per cell at 3 months

SECONDARY OUTCOMES:
Relative change in PCA3 (a prostate cancer-specific gene) expression per cell at 3 months Relative change in prostate volume at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, PhD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Nijmegen, Netherlands